CLINICAL TRIAL: NCT05867381
Title: Slowing Atherothrombosis Progression Through Indoor Air Filtration: A Crossover Trial in Hispanic and Non-Hispanic Adults With Ischemic Heart Disease History
Brief Title: Using Indoor Air Filtration to Slow Atherothrombosis Progression in Adults With Ischemic Heart Disease History
Acronym: SAPIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Duke University (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Zhanghua Chen, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SAPIA_Study; R01ES033707 (NIH)
Record Dates: First submitted 2023-04-23; First posted 2023-05-22 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Air Pollution; Atherosclerosis
Keywords: Air pollution; Particulate matter; Air purifier; HEPA filter; Atherosclerosis; Ischemic Heart Disease; Thrombosis; Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Myocardial Ischemia; Thrombosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A sham filter will be used in the control, to replace HEPA filter in the intervention group. Participants and investigators will be blinded to the intervention type, only investigators who will prepare air filters for intervention will be unblinded for the real air filter type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEPA first and sham (Experimental): This group of participants will be assigned to the intervention of HEPA filtration with the capacity to reduce indoor PM2.5 levels at their residence for 9 months first. After 3-month wash-out period, participants will be assigned to sham filters (air purifier has the same appearance but HEPA filter is removed) for 9 months.
  Interventions: Device: HEPA filtration; Device: Sham filtration
- Sham first and HEPA (Experimental): This group of participants will be assigned to the intervention of sham filtration with HEPA filter removed at their residence for 9 months first. After 3-month wash-out period, participants will be assigned to the HEPA filtration for 9 months.
  Interventions: Device: HEPA filtration; Device: Sham filtration

INTERVENTIONS:
Device: HEPA filtration — HEPA filters with the capacity to reduce PM2.5 levels
Device: Sham filtration — Sham filtration use the same appearance of air purifier but with HEPA filter removed.

SUMMARY:
This double-blind, randomized, crossover trial aims to test the hypothesis that longer-term indoor air filtration intervention can slow atherothrombosis progression by reducing indoor fine particulate matter (PM2.5) exposure in adults with ischemic heart disease history.

DETAILED DESCRIPTION:
This double-blind, randomized, crossover trial will recruit 112 adults with ischemic heart disease history and will investigate potential benefits of indoor high efficiency particulate air (HEPA) filtration on ameliorating the progression of atherothrombosis. Participants will be contacted and recruited to the study based on inclusion and exclusion criteria. After consenting, participants will go through a total of 21-month study period comprised of true HEPA filtration and sham filtration, each of 9-month in duration, and a 3-month wash-out period. After 3-month wash-out period, participants will be switched to the other arm of the intervention. During the trial, project specialists will complete a series of home visits before, in the middle, and after each intervention session to set up air purifiers and indoor and outdoor air pollution monitors, as well as conduct interview to collect questionnaire data, measure vascular function, blood pressure, and collect biospecimens. Participants will self-monitor their daily blood pressure through out the intervention periods. In aim 1, researchers will assess the effect of a 9-month residential HEPA intervention on atherothrombosis progression in 112 participants. In aim 2, the researchers will examine the association between reduction in indoor PM2.5 exposure brought by the intervention and the changes in atherothrombosis progression indicators adjusting for outdoor PM2.5 exposure. In aim 3, researchers will examine atherothrombosis responses (both levels and slopes of change) to the HEPA intervention within four subgroups of participants: 1) non-Hispanics, 2) Hispanics, 3) females, and 4) males.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 84 years old;
* Weight ≥ 110 pounds;
* Nonsmokers for at least 1 year;
* Have ischemic heart disease history, clinically stable for 6 months, without any deterioration in symptoms or episodes of angina based on past electronic medical records;
* Both English and Spanish speaking participants will be included in the recruitment;
* Live in the Los Angeles County.

Exclusion Criteria:

* Have history of degenerative disease of the nervous system such as dementia and Alzheimer's;
* Currently have active cancer treatments;
* The residential house has already had HEPA filters;
* Participants will move out from the current residential address in the next 2 years;
* Participants will spend more than 1 month living outside the primary home;
* Have any health conditions that prohibit collecting health and covariate data and biospecimens;
* Participants' residential houses are not feasible for setting up air purifiers and air pollutants monitors.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | Blood pressure will be monitored daily during each of the 9-month intervention
  Differences between baseline and systolic and diastolic blood pressure measured during and after intervention
Change in carotid-femoral pulse wave velocity | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and carotid-femoral pulse wave velocity measured with Vicorder device during and after intervention
Change in augmentation index | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and augmentation index measured with Vicorder device during and after intervention
Change in von Willebrand factor | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and von Willebrand factor measured during and after intervention
Change in P-selectin | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and P-selectin measured during and after intervention

SECONDARY OUTCOMES:
Change in fasting glucose | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and fasting glucose measured during and after intervention
Change in fasting insulin | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and fasting insulin measured during and after intervention
Changes in lipid profiles | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and low-density lipoprotein, high-density lipoprotein, very-low-density lipoprotein, triglycerides, and total cholesterol levels measured during and after intervention
Change in C-reactive protein | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and C-reactive protein measured during and after intervention
Change in interleukin 6 | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and interleukin 6 measured during and after intervention
Changes in 384 kinds of targeted cardiovascular disease-related proteomic markers | At the baseline, in the middle (4.5 month after intervention) and immediately after each of the 9-month interventions
  Differences between baseline and the relative abundance of 384 kinds of targeted cardiovascular disease-related proteomic markers, such as tumor necrosis factor, E-selectin, intercellular adhesion molecule 1, vascular cell adhesion molecule 1, and leptin, measured with Olink's Explore 384 cardiometabolic panel 1 during and after intervention. The Olink kit is a relative quantification assay and there are no units for the measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanghua Chen, PhD, Principal Investigator — University of Southern California; Junfeng Zhang, PhD, Principal Investigator — Duke University
Locations (1):
- Keck School of Medicine, University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No